CLINICAL TRIAL: NCT01599624
Title: Stress Resilience Training System
Acronym: SRTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency); Perceptronics Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMCSD.2012.0032
Record Dates: First submitted 2012-05-07; First posted 2012-05-16 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Stress; Anxiety; Depression; PTSD
Keywords: Resilience; Perceived stress; PTSD symptoms; Depression; Anxiety; Sleep quality; United States Navy service members
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iPad-based SRTS (Experimental)
  Interventions: Behavioral: Stress Resilience Training System (SRTS)
- iPad-based PMR program (Experimental)
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)

INTERVENTIONS:
Behavioral: Stress Resilience Training System (SRTS) — SRTS training provides both cognitive learning and training in a scientifically-designed stress resilience training approach designed to minimize the adverse effects of stress and also enhance its positive effects. In summary, the SRTS training comprises: (1) Cognitive rules and mental exercises based on expert knowledge and research; (2) Biofeedback stress control exercises based on proven HRV (Heart Rate Variability) algorithms developed by the Institute of HeartMath; and (3) E-Learning presentation of games and simulations to motivate younger trainees. The training is designed to familiarize participants with the iPad and the SRTS program. Participants will be told how to use the system and how often to use the system. SRTS program participants will each be assigned an iPad to take home with them and practice the techniques for a period of two months.
  Arms: iPad-based SRTS
Behavioral: Progressive Muscle Relaxation (PMR) — Progressive muscle relaxation is the systematic tensing and relaxing of 16 different muscle groups, starting with one's toes and ending with one's head (Jacobson, 1938; Conrad & Roth, 2007). PMR users are instructed to inhale as they tense the muscles and exhale as they release the tension. Participants will participate in a two-hour PMR training. PMR participants will be given iPADs with a video recording that guides the user through working each muscle group while instructing them to focus on positive thoughts and feelings and breathing techniques. PMR program participants will each be assigned an iPad to take home with them and practice the techniques for a period of two months.
  Arms: iPad-based PMR program

SUMMARY:
The Stress Resilience Training System (SRTS) program is a stress reduction and resilience building system that blends cognitive training to anticipate the effects of stress with advanced biofeedback to mitigate stress effects and aftereffects, using a game-based learning framework on an iPad platform.

The proposed study will evaluate the effectiveness of the SRTS program at reducing perceived stress, PTSD symptoms, depression, anxiety, sleep quality, coping, attrition and class/operational performance among United States Navy service members.

DETAILED DESCRIPTION:
Military operations and training situations present many physical and psychological challenges for service members to adapt to and overcome. The challenges of these changing conditions necessitate having to cope with stress, which is seen as the negative perceptions, feelings, and emotions that manifest from the subjective physical and/or mental strain on life processes. In addition, service members are returning from deployments having gone through traumatic experiences that can develop into posttraumatic stress disorder (PTSD), depression or other serious conditions.

In an increasing number of military personnel, the adverse effects of service and particularly of stressful combat exposure are significant, long lasting and possibly fatal. Most stress research is focused on treatment, but because stress effects are liable to appear years after exposure, it is imperative that methodologies be developed to mitigate the adverse effects of military-related stress and prevent its post-exposure effects.

It has long been accepted that warfighters adapt to combat stress after the first few experiences and that training can help duplicate this process, with recent studies showing that experienced military personnel are able to control and even utilize stress productively. A key part of what experienced personnel learn is self-awareness of their stress state and self-regulation of stress energy in order to maintain or even improve performance. These skills can be greatly enhanced by combining cognitive learning methodologies grounded in learning theory and biofeedback techniques based on Heart Rate Variability (HRV) with innovative simulation and game-based training tools.

The Stress Resilience Training System (SRTS) program is a stress reduction and resilience building system that blends cognitive training to anticipate the effects of stress with advanced biofeedback to mitigate stress effects and aftereffects, using a game-based learning framework on an iPad platform.

The proposed study will evaluate the effectiveness of the SRTS program at reducing perceived stress, PTSD symptoms, depression, anxiety, sleep quality, coping, attrition and class/operational performance among United States Navy service members.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be Sailors attached to the Training Support Center San Diego (USN).
* All genders and ethnic groups are to be included in the study.

Exclusion Criteria:

* Subjects will be excluded from participation if they will not be at the command for a minimum of 4 months from the start date.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale-10 | baseline, 2 months, 4 months
  This is a 10-item scale designed to measure the degree to which a person perceives aspects of their life as uncontrollable, unpredictable and overwhelming. Participants are asked to indicate how often they have felt a certain way in the last month. The scale utilizes a 5-point likert format with responses ranging from never to very often.
Pittsburgh Sleep Quality Index (PSQI) | baseline, 2 months, 4 months
  The scale consists of seven different components of sleep quality that sum to an overall sleep quality score. A global score of 0-5 indicates good sleep quality while a global score greater than 5 indicates poor sleep quality. The global score as well as the sleep latency and habitual sleep efficiency scores will be used as continuous variables (Buysse, 1989).
Generalized Anxiety Disorder Measure (GAD-7) | baseline, 2 months, 4 months
  The scale was initially developed to screen for generalized anxiety disorder, but has sensitivity and specificity to panic, social anxiety, and PTSD. The instructions ask respondents to indicate how often they have been bothered by problems over the past two weeks. Scores are obtained from likert responses that range from 0 "Not at all" to 4 "Nearly every day". The total score can range from 0 to 21, with scores of 5, 10, and 15 being cutpoints for mild, moderate, and severe anxiety, respectively. The measure will be utilized to gain anxiety symptom severity scores (Spitzer et al., 2006).

SECONDARY OUTCOMES:
PTSD Checklist -Civilian Version (PCL-C) | baseline, 2 months, 4 months
  The PCL is a 17-item self-report measure of the 17 DSM-IV symptoms of PTSD. The PCL has a variety of purposes, including screening individuals for PTSD, diagnosing PTSD and monitoring symptom change during and after treatment. We will use the PCL-C (civilian) version for this study. The PCL-C (civilian) asks about symptoms in relation to "stressful experiences." The PCL-C is useful because it can be used with any population. The symptoms endorsed may not be specific to just one event, which can be helpful when assessing survivors who have symptoms due to multiple events. Typically, it is optimal to assess traumatic event exposure to ensure that a respondent has experienced at least one Criterion A event.
Patient Health Questionnaire (PHQ-9) | baseline, 2 months, 4 months
  The scale measures the severity of depressive symptoms an individual endorses; the range of scores is 0 to 27, with scores of 5, 10, 15, and 20 indicating mild, moderate, moderately severe and severe depression, respectively. The criteria for major depressive disorder (MDD) can be met when a respondent checks "nearly every day" on the first item and checks four of the following items at equal or greater than "more than half the days." The ninth item reflects one's degree of suicidal ideation (SI). We will have a licensed independent practitioner available to whom those with any SI endorsed will be referred for a risk assessment. The PHQ-9 score will be used as a continuous dependent variable (Kroenke et al., 2001).
Response to Stressful Experiences Scale (RSES) | baseline, 2 months, 4 months
  The RSES is a 22-item assessment designed to measure how individuals respond to stress, adversity and trauma. It includes six factors: positive appraisal, spirituality, active coping, self-efficacy, learning and meaning-making and acceptance of limits. Responses for individual questions will be reviewed in addition to the overall score which reflects the strength of the trait (Johnson, 2008).
Brief COPE | baseline, 2 months, 4 months
  The Brief COPE is a 28-item scale designed to measure how people cope with stressful situations. Factor analysis revealed 10 distinct subscales: self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, and planning (Carver, 1997).
Unit Support | baseline, 2 months, 4 months
  The scale measures an individual's perceived degree of cohesion and quality of relationships with other military personnel during a given period of time spent together. Respondents are asked to describe how much they agree or disagree to a number of statements. Scores are obtained on a 5 point likert scale with responses ranging from 1 Strongly disagree to 5 Strongly agree. Higher scores reflect a better quality of relationships and a more unified group (King et al., 2003).
Quality of Life Scale (QOLS) | baseline, 2 months, 4 months
  The QOLS is a 16 item scale assessing quality of life in areas such as physical health, social connections, recreation, etc. (Burckhardt 193).
Performance Indicator | 4 months
  Command-determined performance data will be collected from Training Support Center San Diego.
Attrition Rate | 4 months
  This will be measured as the percentage of service members who drop out of each respective training program. This information will be collected from the command.

OTHER OUTCOMES:
Compliance | end of program (2 or 4 months)
  • For both the SRTS and PMR iPad-based programs, compliance data will be collected and stored on each iPad. Data will include the number of times the program was opened, the date for each session and for how long the program was open on each occasion. Data will be downloaded from iPads when iPads are turned in at the end of two months. • Participants will also be asked to complete a self-report form, indicating how often, on average, they used the program and practiced the techniques per week.

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Johnston, PhD, Principal Investigator — U.S. Navy, Medical Service Corps, Naval Center for Combat & Operational Stress Control (NCCOSC)

IPD SHARING:
Plan to Share IPD: No